CLINICAL TRIAL: NCT03704727
Title: The Effects of Probiotics on Intestinal Permeability in Gastrointestinal Cancer Patients in Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Actial Farmaceutica S.r.l. (Industry); Nutricia, Inc. (Industry)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-18010425
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Intestinal Permeability; Gastrointestinal Irritation; Mucositis
MeSH Terms: conditions — Mucositis | interventions — Probiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- probiotic treatment (Experimental): Probiotic: VSL#3 is a probiotic formula containing a mixture of 9x10^10 CFU/g Lactobacilli strains (Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus casei, and Lactobacillus bulgaricus), 8x10^10 CFU/g Bifidum strains (Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis) and 20x10^10 CFU/g Streptococcus thermophilus. Administred orally
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotics (beneficial microorganisms) VSL#3 is a probiotic formula containing a mixture of 9x10^10 CFU/g Lactobacilli strains (Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus casei, and Lactobacillus bulgaricus), 8x10^10 CFU/g Bifidum strains (Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis) and 20x10^10 CFU/g Streptococcus thermophilus

SUMMARY:
The aim of this study is to test the hypothesis that adjuvant administration of probiotics in cancer patients undergoing chemotherapy can reduce a chemo-induced increased intestinal permeability. Furthermore, we hypothesize that the use of probiotics may reduce the occurrence of gastrointestinal side effects such as diarrhea, abdominal pains, bacterial translocation and infections following chemotherapy.

DETAILED DESCRIPTION:
Treatment of most cancer patients involves radiation and/or chemotherapy which often leads to gastrointestinal toxicity. Cytotoxic chemotherapy in particular often induces several intestinal abnormalities such as mucositis including destruction of intestinal villi, alterations in the gut microbiota, modulation of tight junctions, leading to an increased intestinal permeability. These toxic effects have been observed in several types of chemotherapy and different methods of administering chemotherapy.

The intestinal permeability is regulated and protected by a number factors, including a mucus layer covering the surface of the epithelium. This mucus layer is partly regulated by intestinal bacteria. Therefore it is hypothesized that chemoinduced changes in the intestinal microbiota may possibly affect intestinal permeability. Changes in the intestinal microbiota are seen after only one or a few cycles of chemotherapy treatment in different types of cancers, and could possibly be a contributing factor in the development of mucositis.

It is possible that probiotics may interfere with the ability of pathogenic bacteria to bind to the surface of the intestinal epithelial lining. In vitro studies have shown that probiotics may reduce a post-infective (Escherichia coli) increased intestinal permeability, or increased permeability due to incubation with pro-inflammatory cytokines. VSL#3 is a probiotic formula containing a mixture of 9x10^10 CFU/g Lactobacilli strains (Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus casei, and Lactobacillus bulgaricus), 8x10^10 CFU/g Bifidum strains (Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis) and 20x10^10 CFU/g Streptococcus thermophilus. In vitro and ex vivo studies have suggested that the probiotic bacteria found in VSL#3 may have a reducing effect on intestinal permeability as well as a positive modulating effect on tight junction protein expression. Escherichia coli Nissle 1917 is another bacterial strain that has been shown to be able to mediate the modulation of tight junction proteins and thus intestinal permeability. The precise mechanisms behind the effects of probiotics on intestinal epithelial permeability are not yet clear, but some mechanisms have been proposed, including a reduction in bacterial secretion of proinflammatory cytokines as well as other secreted products from probiotic microbial metabolism.

It is not known whether all probiotic strains exert a similar effect on intestinal permeability, as only very limited clinical research has addressed this relation. However, it is very likely that the specific choice of probiotic bacterial species may play a crucial role. We are only familiar with one clinical trial examining the effect of probiotics on intestinal permeability in adults with cancer undergoing treatment in the form of colectomy, but no adjuvant chemotherapy. Probiotics in the form of Lactobacillus plantarum, Lactobacillus acidophilus and Bifidobacterium longum was administered perioperative and postoperative to patients undergoing colectomy, and the study showed that probiotics improved the integrity of the small intestinal mucosal barrier, induced modulation of the intestinal microbiome as well as a reduction in the postoperative rate of infections.The same researchers also measured serum zonulin in the same subjects, and found that the treatment with probiotics also reduced the concentration of postoperative serum zonulin, and thus inhibited the same increase in intestinal permeability as was the case in the control group.

ELIGIBILITY:
Inclusion Criteria:

* GI cancer (all types) patients undergoing chemotherapy in oncologic department at Rigshospitalet in Copenhagen
* Age >18 years
* Patients with at least three planned chemo therapy sessions left

Exclusion Criteria:

* Pregnant
* Patients who don't speak, write or understand Danish
* Known inflammatory bowel diseases or malabsorption
* Chronic kidney disease (2 x upper limit plasma creatinine)
* Neutropenia (< 1.5 x 109/L neutrophilic granulocytes in peripheral blood)
* Use of antibiotics
* Use of lactulose (laxative) and not able to discontinue three days prior to urin collection (lactulose/mannitol test)
* Use of probiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Intestinal permeability | 4 hours
  Urinary lactulose-mannitol test

SECONDARY OUTCOMES:
Gastrointestinal adverse events | 1 week
  Diarrhea, abdominal pain, abdominal cramps, constipation, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD,MPA, Principal Investigator — University of Copenhagen
Locations (1):
- Departmen of Oncology, Rigshospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No